CLINICAL TRIAL: NCT04599920
Title: Effects of Replacing Red and Processed Meat With Legume-based Foods on Nutrient Intake, Nutritional Status, Food Consumption, and Biomarkers of Cardiovascular Diseases, Colorectal Cancer, and Type 2 Diabetes in Healthy Working Age Men
Brief Title: Effects of Replacing Red Meat With Legumes on Biomarkers of Chronic Diseases in Healthy Men (Leg4Life)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Anne-Maria Pajari, Adjunct Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Leg4Life-HY
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Colorectal Cancer; Cardiovascular Diseases; Type2 Diabetes
Keywords: colorectal cancer; cardiovascular diseases; type2 diabetes; diet; plant protein; animal protein; red meat; legumes
MeSH Terms: conditions — Colorectal Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red meat supplementation providing 25% of protein intake (Active Comparator): A diet supplemented with 760 g of cooked and boneless red meat per week, corresponding the average consumption of red meat in Finnish men.
  Interventions: Dietary Supplement: Partial replacement of red meat with legume-based foods
- Red meat mostly replaced with legume-based foods (Experimental): A diet supplemented with legume-based foods providing 20% of protein intake and with 200 g per week of red meat providing 5% of protein intake.
  Interventions: Dietary Supplement: Partial replacement of red meat with legume-based foods

INTERVENTIONS:
Dietary Supplement: Partial replacement of red meat with legume-based foods — 560 g of cooked and boneless red meat is replaced with legume-based foods providing the equal amount of protein.

SUMMARY:
The aim of this study is to investigate the effects of partial replacement of red meat with legume-based foods on gut metabolism and markers for colorectal cancer as well as markers for cardiovascular diseases and type 2 diabetes in healthy working age men. The study participants will be stratified into two groups with different amounts of red meat in diet: 1) a diet containing 760 g of cooked and boneless red meat, supplying 25% of daily protein intake and 2) a diet supplying 20% of protein intake with legume-based foods and 5% of protein intake with red meat. The participants will get all meat and and legume-based foods from the research center; otherwise they will be asked to follow their habitual diet. Blood, urine, and stool samples will be collected at the baseline and at the end of the 6 week intervention, as well as BMI, blood pressure and body composition. Nutrient intake and food consumption will be analyzed from 4-day food records at the baseline and at the end of the intervention period.

DETAILED DESCRIPTION:
A human intervention study with healthy volunteers will be carried out to investigate the effects of partial replacement of red meat with legume-based foods on gut metabolism and markers for colorectal cancer as well as biomarkers for cardiovascular diseases and type 2 diabetes.

The study will be done in parallel-design, randomized fashion, with healthy male volunteers aged 20-65 years. Inclusion and exclusion criteria are described elsewhere. Duration of the intervention will be 6 weeks.

Intervention groups will be as follows (n=50/group):

Group 1: The habitual diet of participants is supplemented with 760 g of cooked and boneless red meat per week, representing the average meat consumption of Finnish men and supplying 25% of protein intake.

Group 2: The habitual diet of participants is supplemented with legume-based foods providing equal amount of protein as 560 g of red meat and 200 g of red meat per week.

The consumption of red meat and legumes will be kept stable throughout the intervention and participants are advised to avoid consuming any red meat or legumes in addition to those provided from the research center. The investigators also aim to investigate, whether replacing red meat with legumes induces other changes in diet. This information is be important if increasing legume consumption is recommended at the population level.

Before starting the intervention, participants will get dietary advice how to follow their diets. They will get the red meat and legume-based foods for free to help to implement the diets and to enhance compliance.

Blood, urine and fecal samples will be collected at the baseline and at the end of the intervention. Nutrient intake and food consumption during the intervention will be analyzed from 4-day food records at the baseline and at the end. Nutrient intakes will be calculated using a new Finnish 'Aromi' software.

The following data collection and analyses will be carried out at the baseline and at the end of the intervention period:

* height, weight, waist and hip circumferences
* body composition by bioelectrical impedance analysis
* resting blood pressure
* fasting lipid profile in the plasma (total cholesterol, LDL and HDL, triglycerides)
* fasting glucose and insulin, HbA1c in the blood
* high sensitive C-reactive protein
* markers for nutritional status in plasma/serum: hemoglobin, transferrin receptor, ferritin, vitamin B12, folate, vitamin D
* urea/nitrogen in the urine
* total and heme-based N-nitroso compounds in feces, concentrations of bile acids, gut microbiota

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Omnivorous
* No exclusion criteria listed below

Exclusion Criteria:

* Vegan
* Food allergies against ingredients in foods supplemented in the study
* Oral medication for any allergies
* Regular use of food supplements
* Extreme sports
* Inflammatory bowel disease
* Colon irritable
* Coeliac disease
* Any kind of cancer within 5 years
* Continuous antibiotics or less than 3 months of the latest antibiotics use
* Type 1 or 2 diabetes
* Hypercholesterolemia
* Hormonal, liver or kidney disease
* Alcohol consumption more than 24 measures per week
* Smoking, using snuff

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Red meat consumption exceeds the recommendation in 76% of Finnish men, while only 26% of Finnish women eat red meat more than the recommended maximum of 500 g per week. Decreasing meat consumption and replacing meat with legumes would be particularly important and relevant in men.
Enrollment: 100 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the composition of gut microbiota as a measure of modification of dietary protein composition. | 6 weeks
  The composition of gut microbiota is measured using HITChip phylogenetic microarray.
Changes in the concentrations of plasma lipids as a measure of diet modification. | 6 weeks
  The changes in the concentrations of total, LDL, and HDL cholesterol as well as plasma triglycerides.
Changes in the intake of nutrients and nutritional status of participants as a measure of diet modification. | 6 weeks
  The changes in the markers for nutritional status in plasma/serum: hemoglobin, transferrin receptor, ferritin, vitamin B12, folate. The intake of nutrients is calculated from 4-day food records.

SECONDARY OUTCOMES:
Changes in the concentrations of N-nitroso compounds in feces. | 6 weeks
  The changes in gut microbiota are analyzed as a measure of diet modification.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Maria Pajari, PhD, Principal Investigator — University of Helsinki
Locations (1):
- Department of Food and Nutrition, University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
The data collected is confidential and cannot be shared.

REFERENCES:
- [Derived] Back S, Paivarinta E, Pellinen T, Itkonen ST, Lehtovirta M, Erkkola M, Kaartinen NE, Mannisto S, Pajari AM. Nutritional and health benefits of a partial substitution of red and processed meat with non-soy legumes: a 6-week randomized controlled trial in healthy working-age men. Eur J Nutr. 2025 Aug 19;64(6):259. doi: 10.1007/s00394-025-03783-x. PMID 40828321
- [Derived] Itkonen ST, Karhu P, Pellinen T, Lehtovirta M, Kaartinen NE, Mannisto S, Paivarinta E, Pajari AM. Effects of partial replacement of red and processed meat with non-soya legumes on bone and mineral metabolism and amino acid intakes in BeanMan randomised clinical trial. Br J Nutr. 2024 Jan 14;131(1):82-91. doi: 10.1017/S0007114523001514. Epub 2023 Jul 10. PMID 37424311